CLINICAL TRIAL: NCT00168701
Title: Double-Blind, Placebo-Controlled, Dose-Ranging Study to Determine the Efficacy and Safety of BG00012 in Subjects With Relapsing-Remitting Multiple Sclerosis
Brief Title: Efficacy and Safety of BG00012 in MS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-1900
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MRI
MeSH Terms: conditions — Multiple Sclerosis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: BG00012

SUMMARY:
Determine the efficacy, safety, and tolerability of BG00012 in MS patients.

DETAILED DESCRIPTION:
The study will be divided into two parts: Part 1 will be a 24-week, blinded, placebo-controlled treatment phase followed by Part 2, a 24-week blinded, safety extension phase in which all subjects will receive BG00012.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 18 to 55 years old, inclusive, at the time of informed consent.
2. Must have a confirmed diagnosis of relapsing-remitting MS according to McDonald criteria #1-4 (McDonald et al, 2001; Appendix 2).
3. Must have a baseline EDSS between 0.0 and 5.0, inclusive.
4. Must have experienced at least one relapse within the 12 months prior to randomization, with a prior cranial MRI demonstrating lesion(s) consistent with MS OR show evidence of Gd-enhancing lesions of the brain on an MRI performed within the 6 weeks.
5. Male and female subjects must be willing to take appropriate measures to prevent pregnancy.

Exclusion Criteria:

1. Primary progressive, secondary progressive, or progressive relapsing MS (as defined by Lublin and Reingold, 1996 [Appendix 3]).
2. History of malignancy.
3. History of severe allergic or anaphylactic reactions or known drug hypersensitivity.
4. History of abnormal laboratory results indicative of any significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, gastrointestinal, dermatologic, psychiatric, renal, neurologic (other than MS), and/or other major disease.
5. History of human immunodeficiency virus (HIV).
6. History of drug or alcohol abuse (as defined by the Investigator) within the 2 years prior to randomization.
7. An MS relapse that has occurred within the 50 days prior to randomization AND/OR the subject has not stabilized from a previous relapse prior to randomization.
8. Body weight >100 kg.
9. Positive for hepatitis C antibody and/or positive for hepatitis B surface antigen (HBsAg) at screening.
10. Any of the following abnormal blood tests at screening.
11. Any previous treatment with FUMADERM®, FAG-201, or BG00012.
12. A medication history that precludes entry into the study.
13. Female subjects who are currently pregnant or breast-feeding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 260 (Actual)
Dates: Start 2004-10-01 (Actual); Primary Completion 2006-03-31 (Actual); Study Completion 2006-03-31 (Actual)

PRIMARY OUTCOMES:
The primary endpoint for the primary objective is the total number of MRI lesions at Weeks 12, 16, 20, and 24. | Weeks 12, 16, 20, and 24

SECONDARY OUTCOMES:
The secondary endpoints will include measuring the changes in MRIs from baseline until Week 24, changes in other MS measurements q12 weeks, and the annualized relapse rate and proportion of changes at Weeks 24 and 48. | Weeks 24 and 48

CONTACTS AND LOCATIONS:
Overall Officials: Ludwig Kappos, Prof, Principal Investigator — Kantonsspital Basel; Gilmore O'Neill, MB,MRCPI,MMedSc, Study Director — Biogen
Locations (35):
- Czechia (5):
  - Faculty Hospital St. Anne, Bmo
  - Faculty Hospital, Hradec Králové
  - Hospital of Pardubice, Pardupice
  - Faculty Hospital of Plzen, Pilsen
  - General Teaching Hospital, Prague
- Germany (3):
  - Bochum am St. Josef-Hospital, Bochum
  - Heinrich-Heine-Universitat, Düsseldorf
  - George-August-Universitat Goettigen, Goettigen
- Hungary (3):
  - Uzsoki Hospital, Budapest
  - University of Debrecen, Debrecen
  - Petz Aladar County Hospital, Győr
- Netherlands (2):
  - VUMC, Amsterdam
  - Academic Hospital Rotterdam, Rotterdam
- Poland (8):
  - SamodzielnyPubliczny Szpital Kliniczny, Bialystok
  - Niesalezny Zespol Opieki Zdrowognej, Bialystok
  - 10 Wojskowy Szpital Kliniczny z Poliklinika, Bydgoszcz
  - Wojewodzki Szpital Specjalistczny, Gdansk
  - Slaskiej Akademii Medycznej, Katowice-Ligota
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Panstwowy Szpital Kliniczny, Lodz
  - Samodzielny Publiczny Centralny Szpital, Warsaw
- Russia (4):
  - Moscow
  - Novosibirsk
  - Saint Petersburg
  - Veliky Novgorod
- Sweden (2):
  - MS Centrum, Mölndal
  - Karolinska University Hospital, Stockholm
- Kantonsspital Basel, Basel, Switzerland
- Turkey (Türkiye) (3):
  - Hacettepe Unisersitesi, Ankara
  - Istanbul University, Istanbul
  - University of Instanbul, Istanbul
- United Kingdom (4):
  - Multiple Sclerosis Reseach Clinic, London
  - Institute of Neurology, London
  - Royal Hampshire Hospital, Sheffield
  - University Hospital of North Staffordshire, Stoke-on-Trent

REFERENCES:
- [Derived] Mehta D, Miller C, Arnold DL, Bame E, Bar-Or A, Gold R, Hanna J, Kappos L, Liu S, Matta A, Phillips JT, Robertson D, von Hehn CA, Campbell J, Spach K, Yang L, Fox RJ. Effect of dimethyl fumarate on lymphocytes in RRMS: Implications for clinical practice. Neurology. 2019 Apr 9;92(15):e1724-e1738. doi: 10.1212/WNL.0000000000007262. Epub 2019 Mar 27. PMID 30918100
- [Derived] Fox RJ, Kita M, Cohan SL, Henson LJ, Zambrano J, Scannevin RH, O'Gorman J, Novas M, Dawson KT, Phillips JT. BG-12 (dimethyl fumarate): a review of mechanism of action, efficacy, and safety. Curr Med Res Opin. 2014 Feb;30(2):251-62. doi: 10.1185/03007995.2013.849236. Epub 2013 Oct 22. PMID 24131282
- [Derived] Kappos L, Gold R, Miller DH, Macmanus DG, Havrdova E, Limmroth V, Polman CH, Schmierer K, Yousry TA, Yang M, Eraksoy M, Meluzinova E, Rektor I, Dawson KT, Sandrock AW, O'Neill GN; BG-12 Phase IIb Study Investigators. Efficacy and safety of oral fumarate in patients with relapsing-remitting multiple sclerosis: a multicentre, randomised, double-blind, placebo-controlled phase IIb study. Lancet. 2008 Oct 25;372(9648):1463-72. doi: 10.1016/S0140-6736(08)61619-0. PMID 18970976